CLINICAL TRIAL: NCT05108623
Title: A Phase 1, Open-Label Study of the Safety, Tolerability and Preliminary Clinical Activity of Allogeneic Invariant Natural Killer T (iNKT) Cells (agenT-797) as a Single Agent and in Combination With Approved Immune Checkpoint Inhibitors in Patients With Relapsed/ Refractory Solid Tumors
Brief Title: A Study Investigating agenT-797 in Participants With Relapsed/Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MiNK Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1306
Record Dates: First submitted 2021-10-12; First posted 2021-11-05 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Tumor, Solid
Keywords: Tumor; Solid Tumor; Immunotherapy; iNKT cells
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Monotherapy with agenT-797 (Experimental): 3+3 Dose escalation of agenT-797 will be administered as a single intravenous (IV) infusion.
  Interventions: Drug: agenT-797
- Part 2: agenT-797 in Combination with approved ICIs (Experimental): Single prespecified dose of agenT-797 administered by IV infusion in combination with approved ICIs administered in accordance with manufacturer instructions and institutional guidelines as per standard of care
  Interventions: Drug: agenT-797; Drug: Approved ICIs

INTERVENTIONS:
Drug: agenT-797 — agenT-797 is an off-the-shelf cell therapy consisting of ≥ 95% allogeneic human unmodified iNKT cells isolated from 1 healthy donor mononuclear cell apheresis unit and expanded ex vivo.
Drug: Approved ICIs — Nivolumab and pembrolizumab
  Arms: Part 2: agenT-797 in Combination with approved ICIs

SUMMARY:
This is a Phase 1, open-label study to explore the safety, tolerability, and preliminary clinical activity of agenT-797, an unmodified, allogeneic iNKT cell therapy, in participants with relapsed/refractory (r/r) solid tumors, as well as define the recommended phase II dose in solid tumors. This Phase 1 study will also explore the safety, tolerability, and preliminary clinical activity of agenT-797 in combination with approved immune checkpoint inhibitors (ICIs), including pembrolizumab and nivolumab, in participants with r/r solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of relapsed or refractory solid tumor malignancy for which no standard therapy is available or standard therapy has failed
* Measurable disease per RECIST 1.1 as assessed by local site Investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Part 2 only, participants must have progressed per Investigator assessment on pembrolizumab or nivolumab, and agree and are able to continue on the inhibitor(s) while on study
* No other medical, surgical, or psychiatric condition (including active substance abuse) that would interfere with compliance to the protocol, as determined by the Principal Investigator

Exclusion Criteria:

* Concurrent invasive malignancy
* Brain and/or leptomeningeal metastases that are untreated or require current therapy
* Prior radiotherapy within 2 weeks of start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Number Of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline through 12 months
  This will be determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).
Number Of Adverse Events (AEs) By The Dose Of iNKT Cell Therapy | Baseline through 12 months
  This will be determined according to the NCI CTCAE v5.0.
Number Of TEAEs By The Dose Of iNKT Cell Therapy | Baseline through 12 months
  This will be determined according to the NCI CTCAE v5.0.
Severity Grade Of AEs By Dose Of iNKT Cell Therapy | Baseline through 12 months
  This will be determined according to the NCI CTCAE v5.0.
Number Of Dose-limiting Toxicities | Baseline through first 14 days after administration

SECONDARY OUTCOMES:
Persistence Of agenT-797 In Peripheral Blood Samples | Baseline/Day 1 (pre-infusion, 5 minutes, 0.25, 0.5, 1, 2, and 4 hours after cell infusion), and on Days 2, 5, 8, 15, 22, and 29; Weeks 6, 8, and 12; and Months 6, 9, and 12
  This will be measured as a length of time, through collection of peripheral blood mononuclear cells and analysis by flow cytometry.
Objective Response Rate (ORR) | Up to 12 months
  For solid tumors, this will be determined per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 guidelines and for prostate cancer (not evaluable per RECIST 1.1), Prostate Cancer Working Group 3 (PCWG3) will be used.
Duration Of Response (DOR) | Up to 12 months
  For solid tumors, this will be determined per RECIST 1.1 guidelines and for prostate cancer (not evaluable per RECIST 1.1), PCWG3 will be used.
Progression-free Survival (PFS) | Up to 12 months
  For solid tumors, this will be determined per RECIST 1.1 guidelines and for prostate cancer (not evaluable per RECIST 1.1), PCWG3 will be used.
Incidence Of Panel-reactive Antibody | Baseline/Day 1 (pre-infusion), Day 8, Day 15, Day 29, Week 8, Week 12, Month 6, and end of study visit (up to 12 months)
Incidence Of Donor-specific Antibody | Baseline/Day 1 (pre-infusion), Day 8, Day 15, Day 29, Week 8, Week 12, Month 6, and end of study visit (up to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MiNK Therapeutics
Locations (8):
- United States (8):
  - University of Southern California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Norton Cancer Health, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - LifeSpan - Rhode Island Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hadfield MJ, Safran H, Purbhoo MA, Grossman JE, Buell JS, Carneiro BA. Overcoming resistance to programmed cell death protein 1 (PD-1) blockade with allogeneic invariant natural killer T-cells (iNKT). Oncogene. 2024 Mar;43(10):758-762. doi: 10.1038/s41388-024-02948-y. Epub 2024 Jan 29. PMID 38281989
- See also: Nivolumab [Package Insert]. Princeton, NJ: Bristol Myers Squibb Company: 2014. — https://packageinserts.bms.com/pi/pi_opdivo.pdf
- See also: Pembrolizumab [Package Insert]. White House Station, NJ: Merck & Co. Inc.; 2014-2021. — https://www.merck.com/product/usa/pi_circulars/k/keytruda/keytruda_pi.pdf